CLINICAL TRIAL: NCT04573348
Title: Prospective, One Center, Four Groups, Open, Comparative, Controlled Study to Explore T Cells Response to SARS COV 2 Peptides by Metabolic Activity Method in Convalesce and Healthy Individuals Versus Antibody Response
Brief Title: T Cells Response to SARS COV 2 Peptides
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Savicell Diagnostics Ltd (Other)
Responsible Party: Sponsor
Other Study IDs: PBMC _COVID 19
Record Dates: First submitted 2020-09-30; First posted 2020-10-05 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-09

CONDITIONS: Covid19; Corona Virus Infection
Keywords: COV-19; T cells; COV-2 PEPTIDE
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — peripheral Blood samples (27ml) once from each participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Groups 1-4: no intervention will be performed in this study, only blood drawn
  Interventions: Diagnostic Test: Savicell's ImmunoBiopsy™

INTERVENTIONS:
Diagnostic Test: Savicell's ImmunoBiopsy™ — ImmunoBiopsy and ELISA

SUMMARY:
The analysis method described in this protocol is a novel simple plausible immunological approach which is non-invasive, high throughput, real-time quantitative monitoring of metabolic activity (MA) profiles of fresh Peripheral Blood Mononuclear Cells (PBMC) in response to various reagents at different concentrations. The purpose of this study is to evaluate the T cells reactivity to SARS COV 2 immunogenic selected peptides by Metabolic Activity Method in convalesce and healthy individuals and to compare it with Antibody response (ELISA) and clinical information

DETAILED DESCRIPTION:
This is a prospective, four groups, open, comparative, controlled study. A total of 400 completed, evaluated subjects will be enrolled in this study. Main Study Measures: Reactivity of T cells to selected SARS COV-2 peptides by MA test and IgG Antibody response to SARS COV-2 by commercial ELISA test.

Study Procedures:

* Screening
* Informed consent signing
* Medical history review
* Blood collection.
* MA test and ELISA test will be performed at Savicell's Laboratory site.

ELIGIBILITY:
Inclusion Criteria:

* All recruited subjects are between 18 to 90 years old.
* All recruited subjects read the informed consent and then signed the informed consent.
* All recruited subjects filled out the questionnaire form

Exclusion Criteria:

* Subject has active infection or inflammation determined clinically at screening.
* Subject is currently treated with concomitant medication related directly or can affect the immune system as steroids.
* Subject has impaired judgment.
* Known positive HIV, hepatitis B, or hepatitis C, autoimmune disease.
* Known history of a significant medical disorder, which in the investigators' judgment contraindicates the patient's participation.
* Drug or alcohol abuse
* Subject is participating in any other clinical trial for drug investigation within 10 days prior sample collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1 :COVID -19 convalesce individuals that tested positive to COVID -19 by swab PCR test who were severe/acute/moderate - ill with hospitalization/drug treatment/ breathing support and who have passed one months or more since recovering from COVID-19 illness Group 2:Belong to family members who shared a household with donors in group 1 and were exposed at the time of symptomatic disease, without any diagnoses of COVID-19 and tested PCR negative to COVID-19. Group 3:COVID - 19 convalesce individuals that tested positive to COVID -19 by swab PCR test who were mild or asymptomatic and who have passed more than two weeks since recovering from illness. Group 4:COVID - 19 healthy blood donors that keep rules of social distance and wearing a mask.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-05-10 (Estimated); Study Completion 2021-10-10 (Estimated)

PRIMARY OUTCOMES:
Positive and negative diagnosis (scored 0/1 dichotomously) in accordance with test results (MA/ELISA/PCR) | week
  T cells reactivity to SARS COV 2 immunogenic

SECONDARY OUTCOMES:
Prevalence of positive for SARS - COV2 - in healthy donors. | week
  Antibody response (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Shafrira Shai, PhD, Study Director — Savicell Diagnostics Ltd
Locations (1):
- Carmel Medical Center, Haifa, North, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Leslie M. T cells found in coronavirus patients 'bode well' for long-term immunity. Science. 2020 May 22;368(6493):809-810. doi: 10.1126/science.368.6493.809. No abstract available. PMID 32439770
- [Background] Seydoux E, Homad LJ, MacCamy AJ, Parks KR, Hurlburt NK, Jennewein MF, Akins NR, Stuart AB, Wan YH, Feng J, Nelson RE, Singh S, Cohen KW, McElrath MJ, Englund JA, Chu HY, Pancera M, McGuire AT, Stamatatos L. Characterization of neutralizing antibodies from a SARS-CoV-2 infected individual. bioRxiv [Preprint]. 2020 May 12:2020.05.12.091298. doi: 10.1101/2020.05.12.091298. PMID 32511342
- [Background] Robbiani DF, Gaebler C, Muecksch F, Lorenzi JCC, Wang Z, Cho A, Agudelo M, Barnes CO, Gazumyan A, Finkin S, Hagglof T, Oliveira TY, Viant C, Hurley A, Hoffmann HH, Millard KG, Kost RG, Cipolla M, Gordon K, Bianchini F, Chen ST, Ramos V, Patel R, Dizon J, Shimeliovich I, Mendoza P, Hartweger H, Nogueira L, Pack M, Horowitz J, Schmidt F, Weisblum Y, Michailidis E, Ashbrook AW, Waltari E, Pak JE, Huey-Tubman KE, Koranda N, Hoffman PR, West AP Jr, Rice CM, Hatziioannou T, Bjorkman PJ, Bieniasz PD, Caskey M, Nussenzweig MC. Convergent Antibody Responses to SARS-CoV-2 Infection in Convalescent Individuals. bioRxiv [Preprint]. 2020 May 22:2020.05.13.092619. doi: 10.1101/2020.05.13.092619. PMID 32511384